CLINICAL TRIAL: NCT03138707
Title: Demographic Characteristics of Patients Who Die Within Emergency Department
Brief Title: Patients Who Die Within Emergency Department
Status: Completed | Type: Observational
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Umut Gulacti, Principal Investigator, Adiyaman University Research Hospital
Other Study IDs: ADYU 7
Record Dates: First submitted 2017-04-29; First posted 2017-05-03 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Emergencies; Death
MeSH Terms: conditions — Emergencies; Death | interventions — Emergency Service, Hospital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patients who die
  Other Names: patients who die in emergency department

SUMMARY:
Emergency services are a crowded and chaotic environment.

DETAILED DESCRIPTION:
Emergency services are a crowded and chaotic environment. Aim of this study is to investigate the clinic features of emergency patients who die after brought to emergency service.

This retrospective study will be conducted on patients who die within Emergency Department a tertiary hospital over between 01 January 2013 and 31 December 2015.

ELIGIBILITY:
Inclusion Criteria:

* patients who die within emergency department

Exclusion Criteria:

* patients who die outside emergency department patients who die before they were admitted to emergency department

Ages: 0 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients who die within Emergency Department of Adıyaman University Tranining and Research Hospital, between January 01, 2013 and December 31, 2015.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
patients who die within Emergency department | two years
  patients who die by data obtained from medical records

CONTACTS AND LOCATIONS:
Overall Officials: Umut Gulacti, Principal Investigator — Adiyaman University Medical Faculty
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker M, Clancy M. Can mortality rates for patients who die within the emergency department, within 30 days of discharge from the emergency department, or within 30 days of admission from the emergency department be easily measured? Emerg Med J. 2006 Aug;23(8):601-3. doi: 10.1136/emj.2005.028134. PMID 16858089